CLINICAL TRIAL: NCT02230709
Title: IMMEDIATE EFFECTS OF DRY NEEDLING VERSUS DRY NEEDLING AND TENS ON PAIN IN PATIENTS WITH CHRONIC MIOFASCIAL NECK PAIN
Brief Title: Immediate Effects of Dry Needling and Tens in Chronic Neck Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Josue Fernandez Carnero, associate professor, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 50/2012
Record Dates: First submitted 2014-08-28; First posted 2014-09-03 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Myofascial Neck Pain
Keywords: Neck pain; Myofascial pain syndrome; Soreness
MeSH Terms: conditions — Neck Pain; Myofascial Pain Syndromes | interventions — Dry Needling; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dry needling (Experimental): Dry needling treatment on the trigger point number 2 of the trapezius muscle.
  Interventions: Other: Dry Needling
- "TENS" and "dry needling" (Active Comparator): Application of TENS current after dry needling treatment.
  Interventions: Other: "TENS" and "dry needling"

INTERVENTIONS:
Other: Dry Needling — Needling with acupuncture needle in a myofascial trigger point.
  Arms: Dry needling
Other: "TENS" and "dry needling" — Application of TENS current after dry needling technique
  Arms: "TENS" and "dry needling"

SUMMARY:
The aim of this study is to determinate the effects of percutaneous electrical nerve stimulation in the short-term for pain in patients with myofascial chronic neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Neck pain for more than six months of evolution.
* Active Myofascial Trigger Point number 2 on Trapezius muscle.
* Score of more than 2 points in a Visual Analog Scale.

Exclusion Criteria:

* Neck pain specific.
* Radiculopathies.
* Whiplash.
* Dizziness and migraines
* Cervical surgical intervention
* Previous treatment of Dry Needling

Ages: 18 Years to 48 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-11; Primary Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Neck Pain | 4 days
  Visual analog scale. A 100mm VAS, ranging from 0mm (no pain) to 100mm (worst imaginable pain).
Post-needling pain | 4 days
  Visual analog scale. A 100mm VAS, ranging from 0mm (no pain) to 100mm (worst imaginable pain).

SECONDARY OUTCOMES:
Pressure Pain threshold | 4 days
  Pressure needed to evoke pain recognized by patient. Measured using an algometer in Kg/cm2
Range of Motion | 4 days
  The subjects sat in a chair and a CROM goniometer was placed over the head. They were asked to perform active neck movements to the fullest extent of their mobility. Each movement was recorded three times and the average value was calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- CSEU La Salle, Aravaca, Madrid, Spain